CLINICAL TRIAL: NCT05184504
Title: Renal Cell Cancer Registry in Latin American Clinical-phatological Characterization and Outcomes of Renal Cell Carcinoma in Latin America
Brief Title: Clinical-pathological Characterization and Outcomes of Renal Cell Carcinoma in Latin American
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 1120
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pathological diagnosis of renal cell carcinoma: Patients aged 18 years or older, who have been diagnosed with renal cell carcinoma (new case or recurrence) since January 2015 and during the study recruitment period.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.

SUMMARY:
Observational study, retrospective and prospective, of an analytical nature. Data will be collected from medical records and/or through contact with physicians and institutions (secondary data collection). Patients included retrospectively or prospectively will be followed during the data collection period for the evaluation of treatments and survival. No intervention is planned in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age;
* Proven histology of renal cell carcinoma (any subtype);
* Pathological diagnosis of renal cell carcinoma in January 2015 or later and new cases diagnosed during the period of recruitment of each center;
* Have the medical record available and suitable for collecting data on patient characteristics, treatment and outcome.

Exclusion Criteria:

* Synchronous or other primary tumor within the last 3 years (except thyroid cancer or non melanoma skin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older, who have been diagnosed with renal cell carcinoma (new case or recurrence) since January 2015 and during the study recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Build a real-life renal cell cancer database in Brazil and Latin America | 2022

SECONDARY OUTCOMES:
Sociodemographic characteristics checklist | 2022
  Describe sociodemographic characteristics: age at diagnosis, race, education, family income, occupation, personal habits, family history, comorbidities, treatment funding (public or private), treatment institution (public, private or philanthropic).
Clinicopathological characteristics of patients with renal cell cancer checklist | 2022
  date of onset of symptoms, pre-treatment symptoms, histology, clinical and pathological stage, performance status, tests used in staging, date of diagnosis, site of metastases, complications clinics.
Characteristics of systemic treatment checklist | 2022
  date of biopsy; dates, type and lines of drug treatment.
Time between diagnosis and start of treatment. | 2022
  Characteristics of systemic treatment checklist
Causes of delay or discontinuation of each treatment checklist | 2022
  Characteristics of systemic treatment
Progression-free survival in each therapeutic line | 2022
Overall survival | 2022

CONTACTS AND LOCATIONS:
Overall Officials: André Poisl Fay, Principal Investigator — Latin American Cooperative Oncology Group
Locations (16):
- Brazil (16):
  - CINPAM - Centro Integrado de Pesquisa da Amazônia, Manaus, Amazonas
  - Oncocentro Ceará (Rede D'or), Fortaleza, Ceará
  - Hospital Evangélico de Cachoeiro de Itapemirim - Centro de Pesquisas Clínicas em Oncologia (CPCO), Cachoeiro de Itapemirim, Espírito Santo
  - Santa Casa de Misericórdia de Feira de Santana, Feira de Santana, Estado de Bahia
  - NOB - Núcleo de Oncologia da Bahia (Oncoclínicas), Salvador, Estado de Bahia
  - Onco-Vida Instituto Especializado de Oncologia, Brasília, Federal District
  - Hospital do Câncer do Maranhão Dr. Tarquínio Lopes Filho, São Luís, Maranhão
  - Clinica Prognóstica - Centro de Pesquisa Clínica Onconeo, Campo Grande, Mato Grosso do Sul
  - ICTR - Instituto do Câncer e Transplante de Curitiba, Curitiba, Paraná
  - Hospital Napoleão Laureano, João Pessoa, Paraíba
  - Hospital Porto Dias, Belém, Pará
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Clínica de Hematologia e Oncologia Viver, Santa Maria, Rio Grande do Sul
  - CTTB - Centro de Tratamento de Tumores Botafogo (Oncoclínicas), Rio de Janeiro
  - Hemomed Instituto de Oncologia e Hematologia, São Paulo
  - CPO - Centro Paulista de Oncologia (Oncoclínicas), São Paulo

IPD SHARING:
Plan to Share IPD: No